CLINICAL TRIAL: NCT07245550
Title: Thyroid and Adrenal Disorders in ICU Patients With Septic Shock
Brief Title: Thyroid and Adrenal Disorders in ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Radwa mahmoud elsayed, principal investigator, Assiut University
Other Study IDs: TAICU
Record Dates: First submitted 2025-09-26; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Septic Shock
Keywords: septic shock
MeSH Terms: conditions — Shock, Septic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with septic shock in the ICU: Blood sampling for thyroid and adrenal hormones
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood sampling for the hormones

SUMMARY:
A dysregulated host response to infection results in organ failure and sepsis, a potentially fatal illness. Sepsis killed about 11 million people worldwide in 2017 and had a death rate close to 20 %

DETAILED DESCRIPTION:
Sepsis syndromes span a clinical continuum with variable prognoses. Septic shock, the most severe complication of sepsis, carries high mortality. In response to an inciting agent, pro-inflammatory and anti-inflammatory arms of the immune system are activated in concert with the activation of monocytes, macrophages, and neutrophils that interact with the endothelium through pathogen recognition receptors to elaborate cytokines, proteases, kinins, reactive oxygen species, and nitric oxide .Sepsis syndromes caused by multidrug-resistant bacterial strains (methicillin-resistant Staphylococcus, vancomycin-resistant enterococci are on the rise with a current incidence of up to 25%; viruses and parasites cause far fewer cases and are identified in 2% to 4% of cases . It is a well-known fact that the thyroid gland plays an important role in regulating metabolism, growth, and development by secretion of hormones such as thyroxine (T4) and triiodothyronine (T3). In critical illness, changes occur in the hypothalamic-pituitary-thyroid (HPT) axis which leads to euthyroid sick syndrome or non-thyroidal illness syndrome (NTIS). This condition is characterized by decreased T3 levels, normal to low levels of T4, and normal to decreased thyroid-stimulating hormone (TSH) levels despite the absence of intrinsic thyroid disease in patients. The pathophysiology of NTIS involves alterations in thyroid hormone production, peripheral conversion of T4 to T3, and increased degradation of thyroid hormones. During critical illness, cytokines and inflammatory mediators such as tumor necrosis factor-alpha (TNF-α) and interleukin-6 (IL-6) play a significant role in these hormonal changes. Reduced activity of deiodinases, enzymes responsible for the conversion of T4 to T3, further contributes to decreased T3 levels. Critical illness is associated with increased systemic cortisol availability, a vital part of the stress response. Stress can cause life-threatening adrenal crisis when a disease of the hypothalamic-pituitary-adrenal (HPA) axis is present and not adequately treated with stress doses of hydrocortisone. Hence understanding these changes is vital to improve prognosis in patients under intensive care. For instance, in the absence of adrenal insufficiency, stress doses of hydrocortisone can be used to reduce the high vasopressor need in patients suffering from septic shock .In response to stress, adrenal gland generates high levels of glucocorticoid (GC). We call this induced GC (IGC). Unfortunately, 25-60% of septic patients experience relative adrenal insufficiency (RAI). RAI is defined by impaired IGC production in response to stress, which is diagnosed by a delta total cortisol of < 9 μg/dL post-ACTH stimulation. Thus, understanding the endocrine changes and correction of these hormone levels as early as possible may reduce the hospitalization duration, thereby improving the prognosis of the patients. However, there is a lacuna in the literature regarding the level of these hormones at various timelines in critically ill patients classified according to the APACHE II classification in India. With the available data, we aimed to determine the thyroid and cortisol changes in acute severely ill patients and to assess their relationship with the severity of illness.

ELIGIBILITY:
Inclusion criteria

* All Patients who match the diagnostic criteria for sepsis/septic shock as stated
* admitted in ICU

Exclusion Criteria:

1. Patients refuse to be enrolled in the study
2. Patients with previous endocrinal disorders.
3. Patients receiving corticosteroid or thyroid hormonal therapy.
4. Pregnancy or lactation.
5. Previous endocrinal gland surgery.
6. Individuals with pacing rhythms, bundle branch blocks (QRS interval >120 ms),

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with septic shock admitted at intensive care unit and their age is above 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
serum Thyroid and adrenal hormones levels | 24 hours
  measurement of thyroid and adrenal hormones (TSH-FT3-FT4 - cortisol level ) will be measured by ELLISA technique in septic shock patients at ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Radwa m elsayed, MB, Principal Investigator — assuit university hospital
Locations (1):
- Radwa mahmoud, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No